CLINICAL TRIAL: NCT06797479
Title: Detection of Circulating Therapeutic Monoclonal Antibodies in Biological Samples of Gynecological Cancer Patients.
Acronym: IMMUNO_ASSAY
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, SCAMBIA GIOVANNI, Professore, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: ID 7345
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Gynecological Cancer; Immunotherapy
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — To detect the ICI mAbs in patients' blood plasma samples, we select three anti PD-1 mAbs (cemiplimab, dostarlimab and pembrolizumab) as prognostic biomarkers which will be quantified using different biochemical/analytical assays.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Blood samples for the analysis of sildenafil in plasma — To detect the ICI mAbs in patients' blood plasma samples, we select three anti PD-1 mAbs (cemiplimab, dostarlimab and pembrolizumab) as prognostic biomarkers which will be quantified using different biochemical/analytical assays.

SUMMARY:
Quantification of anti PD-1 mAbs in cancer patients is extremely important to monitor pharmacokinetics and effectiveness of immunotherapy. To detect the ICI mAbs in patients' blood plasma samples, we select three anti PD-1 mAbs (cemiplimab, dostarlimab and pembrolizumab) as prognostic biomarkers which will be quantified using different biochemical/analytical assays.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of gynecological malignancy;
* Patients currently undergoing or scheduled to undergo immunotherapy as part of their treatment regimen;
* Age > 18 years;
* Patients who are able and willing to provide written informed consent to participate in the study.
* Availability of biological samples.

Exclusion Criteria:

* Patients receiving concurrent treatment with other investigational drugs or therapies that may interfere with immunotherapy.
* Presence of significant comorbidities or other medical conditions that, in the opinion of the investigator, would interfere with study participation or interpretation of results (e.g., severe autoimmune diseases, uncontrolled infections);
* Pregnant or breastfeeding women;
* Patients who have received prior monoclonal antibody therapy that could affect the study results;
* Patients who are unable or unwilling to comply with the study procedures and follow-up requirements;
* Brain metastases;
* History of other malignancies within the last 5 years, except for adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gynecological cancers undergoing immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Quantification of anti PD-1. | From enrollment to the end of treatment at 4 weeks
  Quantification of anti PD-1 mAbs in cancer patients is extremely important to monitor pharmacokinetics and effectiveness of immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS